CLINICAL TRIAL: NCT04428528
Title: Pilot Study to Evaluate Photoacoustic Imaging for Characterizing Breast Masses and Breast Tumor Response to Neoadjuvant Chemotherapy
Brief Title: Photoacoustic Imaging for Characterizing Breast Masses and Breast Tumor Response to Neoadjuvant Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Radiation Oncologist and Clinical Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 456-2016
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: chemotherapy; photoacoustic imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant Chemotherapy Monitoring: The first arm Neoadjuvant Chemotherapy Monitoring will investigate changes of measured photoacoustic markers and compare to these to histopathological indicators of breast tumor response to NAC. Changes in photoacoustic parameters will be made to a pre-treatment point over the course of treatment. Treatment will not be modified on the basis of our observations.
  in this pilot observational study
  Interventions: Device: Photoacoustics Imaging System
- Breast Mass Characterization: The second arm Breast Mass Characterization will investigate if breast masses (benign vs. malignant) can be characterized during clinical diagnostic work-up. Differences in the photoacoustic tissue-properties will be compared to histopathological evaluation.
  Interventions: Device: Photoacoustics Imaging System

INTERVENTIONS:
Device: Photoacoustics Imaging System — Characterizing breast masses for photoacoustic markers measurements

SUMMARY:
Our objective in this pilot study will be to identify PA parameters that can distinguish benign vs. malignant lesions, and also, if PA parameters change with within breast tumors during chemotherapy treatment over time.

DETAILED DESCRIPTION:
This study will investigate photoacoustic tissue characteristics of breast lesions both at diagnosis, and within a separate subgroup of patients, physiological changes in breast tumors during neoadjuvant chemotherapy (NAC). Our objective in this pilot study will be to identify PA parameters that can distinguish benign vs. malignant lesions, and also, if PA parameters change with within breast tumors during chemotherapy treatment over time. Our hope is to use this information to correlate with pathological response.

ELIGIBILITY:
Cohort 1 - Neoadjuvant Chemotherapy Monitoring:

Inclusion Criteria:

* Subjects must give appropriate written informed consent prior to participation in the study;
* Subjects must be able and willing to comply with the safety procedures during the Scanning Period;
* Subjects must be men and women of between 20 to 80 years of age, inclusive, on the day the Informed Consent Form is signed;
* Subjects must be receiving neoadjuvant chemotherapy for locally-advanced breast cancer.
* Biopsy-confirmed diagnosis of locally advanced breast cancer; of all molecular subtypes (ER+/-, PR+/-, HER2+/-).

Exclusion Criteria:

* Subjects with a past medical history of abnormalities, significant injury, or medical or surgical procedures (e.g. Silicone/saline implants) involving either breast, exclusive of the lesion at issue;
* Subjects with any dermatologic abnormalities (including tattoos, open sores, or breached skin) involving either breast;
* Subjects with a current or past medical history of connective tissue disease;
* Subjects who are pregnant or lactating;
* Subjects with an implanted electronic device such as a cardiac pacemaker, defibrillator, or neurological stimulator;
* Subjects with a history or expectation of significant anxiety associated with undergoing diagnostic evaluations;
* Subjects with a history of musculoskeletal disease which may predispose them to discomfort during the Scanning Period;
* Subjects with a known sensitivity to low-power infrared radiation (e.g., as a result of a dermatologic condition); and
* Subjects, who, in the opinion of the investigator or clinical research coordinator, may not otherwise be appropriate for inclusion into the study.

Cohort 2 - Breast Mass Characterization:

Inclusion Criteria:

* Subjects must give appropriate written informed consent prior to participation in the study;
* Subjects must be able and willing to comply with the safety procedures during the Scanning Period;
* Subjects must be men and women of between 20 to 80 years of age, inclusive, on the day the Informed Consent Form is signed;
* Subjects must be referred to breast diagnostic clinic for investigation of a breast mass.

Exclusion Criteria:

* Subjects with a past medical history of abnormalities, significant injury, or medical or surgical procedures (e.g.,silicone/saline implants) involving either breast, exclusive of the lesion at issue;
* Subjects with any dermatologic abnormalities (including tattoos, open sores, or breached skin) involving either breast;
* Subjects with a current or past medical history of connective tissue disease;
* Subjects who are pregnant or lactating;
* Subjects with an implanted electronic device such as a cardiac pacemaker, defibrillator, or neurological stimulator;
* Subjects with a history or expectation of significant anxiety associated with undergoing diagnostic evaluations;
* Subjects with a history of musculoskeletal disease which may predispose them to discomfort during the Scanning Period;
* Subjects with a known sensitivity to low-power infrared radiation (e.g., as a result of a dermatologic condition); and
* Subjects, who, in the opinion of the investigator or clinical research coordinator, may not otherwise be appropriate for inclusion into the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort 1 - Neoadjuvant Chemotherapy Monitoring:
  Men and women with either a biopsy confirmed diagnosis of breast cancer and receiving neoadjuvant chemotherapy.
  Cohort 2 - Breast Mass Characterization:
  Men and women suspected of having a mammary, benign or malignant mass and are schedule to undergo diagnostic and clinical work-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2025-02-13 (Estimated); Study Completion 2029-02-13 (Estimated)

PRIMARY OUTCOMES:
Treatment response correlation between photoacoustic parameters and histopathological measurement. | 4 to 8 months
  The primary study endpoint will investigate changes of measured photoacoustic markers and compare to these to histopathological indicators of breast tumor response to NAC. Changes in photoacoustic parameters (hemoglobin concentration, oxygen saturation, tumor structure) will be made to a pre-treatment point over the course of treatment. Treatment will not be modified on the basis of our observations in this pilot observational study.

SECONDARY OUTCOMES:
Breast mass characterization | 30 days
  The secondary study endpoint will investigate if breast masses (benign vs. malignant) can be characterized by PA during clinical diagnostic work-up. Differences in the photoacoustic tissue-properties will be compared to histopathological evaluation. No diagnostic information from PA measurements will be used for patient-care/diagnosis as a result of our observations in this pilot observational study

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Czarnota, PhD, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada